CLINICAL TRIAL: NCT07090109
Title: Partnering to Impact Testing in the Commonwealth for Hereditary Cancers (PITCH)
Brief Title: PITCH - Impacting Hereditary Cancer Testing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rachel Miller (Other)
Responsible Party: Sponsor-Investigator, Rachel Miller, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 98088
Record Dates: First submitted 2025-07-22; First posted 2025-07-29 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Cancer; Genetic Testing; Genetic Counseling
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Educational Video (Experimental): Participants will complete a survey before and after viewing an educational video
  Interventions: Behavioral: Genetic testing education video

INTERVENTIONS:
Behavioral: Genetic testing education video — patient education video about genetic testing for hereditary cancers

SUMMARY:
The goal of this clinical trial is to assess patients' knowledge and attitudes about genetic testing before and after viewing an educational video. The main questions it aims to answer are:

* Did the video change participants' knowledge and attitudes about genetic testing?
* Did participants make an informed choice about pursuing genetic testing?

Participants will:

* Complete a baseline survey
* View educational video
* Complete follow-up survey

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with a cancer that can be associated with hereditary forms of cancer

Exclusion Criteria:

* previously undergone multi-gene panel testing for hereditary cancers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Multi-Dimensional Measure of Informed Choice (MMIC) - Cancer Knowledge Scale | Baseline and post intervention (approximately 30 minutes)
  The MMIC is a compound assessment tool with three elements which are used together to differentiate an informed choice from a less informed choice. An informed choice is demonstrated by: Achieving =75% (6 of 8 questions) correct responses on the knowledge scale AND Making a decision that is in keeping with one's values related to the outcome (positive vs. negative) A less informed choice is demonstrated by: Achieving <75% correct responses on the knowledge scale OR Achieving =75% correct responses on the knowledge scale but making a decision that is inconsistent with one's values (e.g., a patient values the information that may be obtained but chose not to undergo testing OR a patient does not value the information and chose to undergo testing)

SECONDARY OUTCOMES:
Number of participants completing genetic testing | 90 days
  Number of participants that complete testing after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Miller, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States